CLINICAL TRIAL: NCT06057428
Title: Activity Levels Amongst Elderly Patients with Symptomatic Lumbar Spinal Stenosis Before and After Decompressive Surgery
Brief Title: Activity Levels Amongst Patients with Lumbar Spinal Stenosis
Acronym: B-ATLAS
Status: Recruiting | Type: Observational
Sponsor: Region Zealand (Other)
Collaborators: Region Syddanmark (Other)
Responsible Party: Principal Investigator, Oliver Bremerskov Zielinski, Principal Investigator, Region Zealand
Other Study IDs: B-ATLAS2; 010-0194/22-3000 (Registry Identifier: B-ATLAS)
Record Dates: First submitted 2023-09-11; First posted 2023-09-28 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Lumbar Spinal Stenosis
Keywords: Spinal stenosis; Elderly; Activity; Surgery
MeSH Terms: conditions — Spinal Stenosis; Motor Activity

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with lumbar spinal stenosis: Patients diagnosed with lumbar spinal stenosis and referred to operation. Measurements of activity levels will be undertaken before operation, and compared to after operation.
  Interventions: Procedure: Decompressive surgery

INTERVENTIONS:
Procedure: Decompressive surgery — Decompressive surgery for lumbar spinal stenosis

SUMMARY:
Lumbar spinal stenosis (LSS) is one of the most common degenerative diseases of the spinal column, with symptoms including low back pain which worsens with ambulation, poor balance, decreased activity due to pain, and a marked decrease in quality of life (QoL). Prevalence rises with age, and current treatment options range from varied conservative management strategies, to surgical intervention with decompression of neural structures.

While the effects of surgical decompression on back pain and QoL has been widely researched, the effects of surgery on activity levels is less well understood. Though patients generally have subjective improvements in this parameter after surgery, objective measurements in this patient group have been lacking.

This study aims to investigate the effects of decompressive surgery on activity levels in elderly patients with LSS. Measurements of activity will be taken before and after decompressive surgery, as well as with regular intervals during a two-year follow-up period.

A better understanding of the effect that LSS has on activity may lead to more patients being able to receive surgical treatment, which is hypothesized to lead to an increase in QoL and less perceived disability amongst this patient group.

DETAILED DESCRIPTION:
Disease background:

While lumbar spinal stenosis (LSS) is one of the most common degenerative diseases of the spinal column, there is no universally accepted definition of LSS, and no accepted radiologic diagnostic criteria. LSS most often refers to a narrowing in the central canal of the vertebrae, the lateral recess, or the neural foramen. Changes to these can occur due to acquired degenerative spondylosis or spondylolisthesis, or more rarely due to conditions such as ankylosing spondylitis and space-occupying lesions, or congenital abnormalities. LSS can be classified according to anatomical location, etiology or severity of narrowing, though no validated classification has been published.

The lack of concrete definition has caused difficulties in estimating the prevalence of LSS. Studies using community-based sampling has shown a prevalence of acquired LSS, defined as a narrowing of the central canal to ≤ 10mm in the anterior-posterior (AP) direction, of 7.3%. The prevalence has been shown to rise with age, from 4.0% affected at < 40 years of age, to 14.3% amongst patients ≥ 60. No significant differences have been observed in overall prevalence according to gender, although there seems to be a slightly higher prevalence amongst elderly females than males.

Although LSS is often asymptomatic, common symptoms of LSS include low back pain, which worsens with prolonged ambulation, lumbar extension and standing, and which is relieved by rest and forward flexion, as well as lumbar radiculopathy. Patients may also complain of poor balance, and physical examination findings may include a wide-based gait and abnormal Romberg results. Symptoms are thought to occur due to compression of microvascular structures in the nerves, allowing for neural ischemia and defects in nerve conduction, and venous pooling resulting in inadequate oxygenation and metabolite accumulation.

Current treatment options for LSS range across both conservative and surgical management strategies. Conservative management has traditionally been regarded as first-line treatment, with a combination approach of physical therapy and pharmacological treatment with NSAIDs and analgesics. Epidural steroid injections have been used for symptom management, though with limited short and long-term benefits. Surgical management is often indicated in patients with ongoing pain despite attempts at conservative management for 3-6 months. Choice of surgical strategy to relieve the pressure on the neural structures depends on the anatomical location of stenosis and number of stenotic segments, as well as the intraoperative assessment of stability.

The effect of surgical decompression on disability, leg pain and back pain has been widely evaluated, but studies of the effect on postural control are sparse. The present study aims to investigate the effect of surgical decompression of symptomatic lumbar spinal stenosis on postural control by assessment of sway measures before and after surgery.

Activity levels:

Physical activity (PA) has been demonstrated to be correlated to physical and mental wellbeing, having been shown to offer significant benefits including preventing and managing cardiovascular disease, cancer, and diabetes, as well as reducing symptoms of depression and anxiety. A dose-response relationship has been observed, and while all PA can be beneficial, higher levels can have more positive effects. Likewise, the negative consequences of sedentary behaviour are well established, hereunder increasing risks of metabolic and musculoskeletal disorders as well as all-cause mortality. As such, PA as both an intervention tool and as a measurement of effect has been becoming increasingly prevalent in the literature.

It is currently recommended that adults should undertake regular PA, with a minimum of 150-300 min of moderate-vigorous physical activity (MVPA) every week. Adults who do not achieve this can be classified as physically inactive. It is worth keeping in mind though, that no definition of MVPA exists, as such a definition would need to be highly individualized.

Efforts have been made to quantify PA in the context of research; the doubly labelled water (DLW) technique has been shown to be highly accurate in measuring total daily energy expenditure and is considered the gold standard when measuring activity levels. However, as this technique is expensive, time-intensive and imposes a high degree of subject interference, it is not practical for large-scale studies.

Other measurements of activity have been developed and validated, including self-report questionnaires, self-report activity diaries, direct observation, and the use of devices such as accelerometers, pedometers, heart-rate monitors, and armbands. Among these, the use of accelerometers as an activity monitoring device has become increasingly prevalent due to the high frequency of measurements, large memory capacity, low subject interference and ability to differentiate between differing levels of activity. Accelerometer use has likewise been recommended as a clinical measurement of PA when undertaking intervention studies and has seen a rise in use in the field of orthopaedics.

Patients with LSS are often classified as physically inactive due to the ambulatory limitations that symptomatic LSS can present with, and rarely meet the abovementioned recommendations for PA, despite evidence suggesting the benefits of PA for LSS patients. Previous studies have not been able to prove a significant effect of decompressive surgery on activity levels for LSS patients six months post-operatively, measured by accelerometer. However, while comparable studies on patients undergoing total hip arthroplasty likewise found no significant improvement in activity levels after six months, studies with longer follow-up, up to a year post-operatively, have been able to show an activity level comparable to healthy control individuals. Likewise, studies measuring activity levels on LSS patients undergoing decompressive surgery using pedometer readings have been able to show a significant increase in activity after 12 months.

Activity monitoring device:

The ActiGraph wGT3X-BT is a triaxial accelerometer, recording inertia in three planes at a sampling rate up to 100 Hz. A proprietary filter can be applied to eliminate artifacts due to movement not caused by human activity, and data is summed as a total activity count per minute, which can then be used to estimate PAEE and MVPA. The wGT3X-BT has been widely validated against gold standard measurements such as DLW, and in appropriate patient groups such as the elderly, and has been shown to be valid and reliable in assessing physical activity intensity.

Rationale of the study:

This study will be the first to correlate the effects of decompressive surgery in patients with symptomatic LSS with activity levels, and associated quality of life increases. Previous studies have been hampered by low power due to sampling size limitations, and short follow-up regimes, both of which this study seeks to manage through multi-centre collaboration and inclusion, and a follow-up regime spanning two years from the time of surgery.

It is expected that the results of our study can facilitate an increased understanding of the role of activity when considering surgical management of symptomatic LSS patients, as well as enable targeted treatment of patients with LSS.

Research question:

Do elderly patients with symptomatic LSS, who have undergone decompressive surgery, show an improvement in activity level compared to pre-operative values?

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Referred to decompressive spinal surgery due to symptomatic lumbar spinal stenosis at ≥ 1 level
* Central canal LSS grade B or C (Schizas classification) at ≥ 1 level by Magnetic Resonance Imaging
* Minimum of 3 months of unsuccessful non-operative treatment

Exclusion Criteria:

* Signs of malignancy or infection in the spinal column
* Severe comorbidities incl. neurodegenerative conditions which may contribute to balance problems
* Revision surgery (previous decompression surgery at the same vertebral level)
* Spinal surgery up to 1 year prior to the date of inclusion
* Mini Mental State Exam (MMSE) score of ≤ 27 points
* Degenerative spondylolisthesis more than 3mm on pre-operative imaging diagnostics

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients over 65 years of age referred to decompressive surgery for lumbar spinal stenosis
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Activity level | Before surgery and 3, 6, 12 and 24 months after surgery
  Activity level, measured by total activity counts per day (TAC/d)

SECONDARY OUTCOMES:
Physical activity | Before surgery and 3, 6, 12 and 24 months after surgery
  Physical activity, measured by time spent in MVPA (minutes/day)
Physical activity | Before surgery and 3, 6, 12 and 24 months after surgery
  Physical activity, measured by physical activity energy expenditure (PAEE) (Kilojoules/d)
Physical inactivity | Before surgery and 3, 6, 12 and 24 months after surgery
  Physical inactivity, measured by sedentary time (hours/d)
Quality of life | Before surgery and 3, 6, 12 and 24 months after surgery
  Subjective QoL, measured by European Quality of Life - 5 Dimensions score (EQ-5D) The EQ-5D consists of six questions regarding current perceived health status and quality of life.
  Questions 1 - 5 have a range of 1 to 3, lower is better. The answer to questions 6 is given on a scale of 0 to 100, where lower is better.
Functional disability | Before surgery and 3, 6, 12 and 24 months after surgery
  Subjective functional disability, measured by Zurich Claudication Questionnaire score (ZCQ) The ZCQ consists of 12 questions for all patients, and a further six questions for patients who have received treatment.
  The questionnaire is divided into three subscales:
  Symptom severity scale (questions 1 - 7): range of the score is 1 to 5, lower is better.
  Physical function scale (questions 8 - 12): range of the score is 1 to 4, lower is better.
  Satisfaction with treatment scale (questions 13 - 18): range of the score is 1 to 4, lower is better.
Self-reported activity | Before surgery and 3, 6, 12 and 24 months after surgery
  Self-reported activity, measured by International Physical Activity Questionnaire - Short Form score (IPAQ-SF) The IPAQ-SF is a short form health survey consisting of 4 questions relating to self-reported physical activity during the last week.
  Each question asks the participant to note how many days during the past week that they carried out vigorous, moderate, light, or sedentary activity. If the number of days is greater or equal to 1, the participant is asked to estimate the amount of hours and minutes they have spent doing that activity.
Quality of life | Before surgery and 3, 6, 12 and 24 months after surgery
  Subjective Quality-of-life, measured by the Short Form Health Survey (SF-36). The SF-36 is a short form questionnaire concerning patients perceived health and quality-of-life (QoL). It consists of 36 questions regarding various aspects of the patients health status, including current and past perceived physical and mental health, and subjective physical function.
  Questions 1,2 and 20 - 22 each have a range of 1 to 5, lower is better. Question 32 likewise has a range of 1 - 5, though where higher is better. Questions 3 - 12 have a range of 1 - 3, higher is better. Questions 13 - 19 have a range of 1 - 2, higher is better. Questions 23 - 31 and 33 - 36 have a range of 1 - 5. The better score depends on the specific question.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver B Zielinski, MD, Principal Investigator — Orthopaedic Department, Zealand University Hospital
Locations (2):
- Denmark (2):
  - Ortopædkirurgisk afdeling, Sjællands Universitetshospital Køge, Køge
  - Rygcenter Syddanmark, Middelfart Sygehus, Middelfart

IPD SHARING:
Plan to Share IPD: Yes
All deidentified individual participant data collected during the trial will be made available to researchers who provide a methodologically sound proposal for use, subject to approval by the study authors.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: A deidentified copy of all individual participant data will be kept by the authors of the study for 10 years following study end. After this time period, the full data set will be archived by the Danish National Archives with no planned end date.
Access Criteria: Reasonable request for access can be made by writing to ozi@regionsjaelland.dk or rudb@regionsjaelland.dk in a time period consisting of 10 years after study end. After this period, requests for access can be made to the Danish National Archives at data@sa.dk.

REFERENCES:
- [Background] Binder DK, Schmidt MH, Weinstein PR. Lumbar spinal stenosis. Semin Neurol. 2002 Jun;22(2):157-66. doi: 10.1055/s-2002-36539. PMID 12524561
- [Background] Schroeder GD, Kurd MF, Vaccaro AR. Lumbar Spinal Stenosis: How Is It Classified? J Am Acad Orthop Surg. 2016 Dec;24(12):843-852. doi: 10.5435/JAAOS-D-15-00034. PMID 27849674
- [Background] Yabuki S, Fukumori N, Takegami M, Onishi Y, Otani K, Sekiguchi M, Wakita T, Kikuchi S, Fukuhara S, Konno S. Prevalence of lumbar spinal stenosis, using the diagnostic support tool, and correlated factors in Japan: a population-based study. J Orthop Sci. 2013 Nov;18(6):893-900. doi: 10.1007/s00776-013-0455-5. Epub 2013 Aug 21. PMID 23963588
- [Background] Katz JN, Dalgas M, Stucki G, Katz NP, Bayley J, Fossel AH, Chang LC, Lipson SJ. Degenerative lumbar spinal stenosis. Diagnostic value of the history and physical examination. Arthritis Rheum. 1995 Sep;38(9):1236-41. doi: 10.1002/art.1780380910. PMID 7575718
- [Background] Lurie J, Tomkins-Lane C. Management of lumbar spinal stenosis. BMJ. 2016 Jan 4;352:h6234. doi: 10.1136/bmj.h6234. PMID 26727925
- [Background] Lee BH, Moon SH, Suk KS, Kim HS, Yang JH, Lee HM. Lumbar Spinal Stenosis: Pathophysiology and Treatment Principle: A Narrative Review. Asian Spine J. 2020 Oct;14(5):682-693. doi: 10.31616/asj.2020.0472. Epub 2020 Oct 14. PMID 33108834
- [Background] Mazanec DJ, Podichetty VK, Hsia A. Lumbar canal stenosis: start with nonsurgical therapy. Cleve Clin J Med. 2002 Nov;69(11):909-17. doi: 10.3949/ccjm.69.11.909. PMID 12430977
- [Background] Liu K, Liu P, Liu R, Wu X, Cai M. Steroid for epidural injection in spinal stenosis: a systematic review and meta-analysis. Drug Des Devel Ther. 2015 Jan 30;9:707-16. doi: 10.2147/DDDT.S78070. eCollection 2015. PMID 25678775
- [Background] Kovacs FM, Urrutia G, Alarcon JD. Surgery versus conservative treatment for symptomatic lumbar spinal stenosis: a systematic review of randomized controlled trials. Spine (Phila Pa 1976). 2011 Sep 15;36(20):E1335-51. doi: 10.1097/BRS.0b013e31820c97b1. PMID 21311394
- [Background] Sengupta DK, Herkowitz HN. Lumbar spinal stenosis. Treatment strategies and indications for surgery. Orthop Clin North Am. 2003 Apr;34(2):281-95. doi: 10.1016/s0030-5898(02)00069-x. PMID 12914268
- [Background] Aadahl M, Kjaer M, Jorgensen T. Associations between overall physical activity level and cardiovascular risk factors in an adult population. Eur J Epidemiol. 2007;22(6):369-78. doi: 10.1007/s10654-006-9100-3. Epub 2007 Feb 28. PMID 17333472
- [Background] Park JH, Moon JH, Kim HJ, Kong MH, Oh YH. Sedentary Lifestyle: Overview of Updated Evidence of Potential Health Risks. Korean J Fam Med. 2020 Nov;41(6):365-373. doi: 10.4082/kjfm.20.0165. Epub 2020 Nov 19. PMID 33242381
- [Background] Bull FC, Al-Ansari SS, Biddle S, Borodulin K, Buman MP, Cardon G, Carty C, Chaput JP, Chastin S, Chou R, Dempsey PC, DiPietro L, Ekelund U, Firth J, Friedenreich CM, Garcia L, Gichu M, Jago R, Katzmarzyk PT, Lambert E, Leitzmann M, Milton K, Ortega FB, Ranasinghe C, Stamatakis E, Tiedemann A, Troiano RP, van der Ploeg HP, Wari V, Willumsen JF. World Health Organization 2020 guidelines on physical activity and sedentary behaviour. Br J Sports Med. 2020 Dec;54(24):1451-1462. doi: 10.1136/bjsports-2020-102955. PMID 33239350
- [Background] Tremblay MS, Aubert S, Barnes JD, Saunders TJ, Carson V, Latimer-Cheung AE, Chastin SFM, Altenburg TM, Chinapaw MJM; SBRN Terminology Consensus Project Participants. Sedentary Behavior Research Network (SBRN) - Terminology Consensus Project process and outcome. Int J Behav Nutr Phys Act. 2017 Jun 10;14(1):75. doi: 10.1186/s12966-017-0525-8. PMID 28599680
- [Background] MacIntosh BR, Murias JM, Keir DA, Weir JM. What Is Moderate to Vigorous Exercise Intensity? Front Physiol. 2021 Sep 22;12:682233. doi: 10.3389/fphys.2021.682233. eCollection 2021. PMID 34630133
- [Background] Melanson EL Jr, Freedson PS. Physical activity assessment: a review of methods. Crit Rev Food Sci Nutr. 1996 May;36(5):385-96. doi: 10.1080/10408399609527732. PMID 8725670
- [Background] Westerterp KR. Assessment of physical activity: a critical appraisal. Eur J Appl Physiol. 2009 Apr;105(6):823-8. doi: 10.1007/s00421-009-1000-2. Epub 2009 Feb 11. PMID 19205725
- [Background] Sylvia LG, Bernstein EE, Hubbard JL, Keating L, Anderson EJ. Practical guide to measuring physical activity. J Acad Nutr Diet. 2014 Feb;114(2):199-208. doi: 10.1016/j.jand.2013.09.018. Epub 2013 Nov 28. No abstract available. PMID 24290836
- [Background] Sliepen M, Lipperts M, Tjur M, Mechlenburg I. Use of accelerometer-based activity monitoring in orthopaedics: benefits, impact and practical considerations. EFORT Open Rev. 2020 Jan 28;4(12):678-685. doi: 10.1302/2058-5241.4.180041. eCollection 2019 Dec. PMID 32010456
- [Background] Norden J, Smuck M, Sinha A, Hu R, Tomkins-Lane C. Objective measurement of free-living physical activity (performance) in lumbar spinal stenosis: are physical activity guidelines being met? Spine J. 2017 Jan;17(1):26-33. doi: 10.1016/j.spinee.2016.10.016. Epub 2016 Oct 25. PMID 27793759
- [Background] Smuck M, Muaremi A, Zheng P, Norden J, Sinha A, Hu R, Tomkins-Lane C. Objective measurement of function following lumbar spinal stenosis decompression reveals improved functional capacity with stagnant real-life physical activity. Spine J. 2018 Jan;18(1):15-21. doi: 10.1016/j.spinee.2017.08.262. Epub 2017 Sep 28. PMID 28962914
- [Background] Harding P, Holland AE, Delany C, Hinman RS. Do activity levels increase after total hip and knee arthroplasty? Clin Orthop Relat Res. 2014 May;472(5):1502-11. doi: 10.1007/s11999-013-3427-3. Epub 2013 Dec 19. PMID 24353051
- [Background] von Rottkay E, Rackwitz L, Rudert M, Noth U, Reichert JC. Function and activity after minimally invasive total hip arthroplasty compared to a healthy population. Int Orthop. 2018 Feb;42(2):297-302. doi: 10.1007/s00264-017-3541-z. Epub 2017 Jul 12. PMID 28702750
- [Background] Schulte TL, Schubert T, Winter C, Brandes M, Hackenberg L, Wassmann H, Liem D, Rosenbaum D, Bullmann V. Step activity monitoring in lumbar stenosis patients undergoing decompressive surgery. Eur Spine J. 2010 Nov;19(11):1855-64. doi: 10.1007/s00586-010-1324-y. Epub 2010 Feb 26. PMID 20186442
- [Background] Chomistek AK, Yuan C, Matthews CE, Troiano RP, Bowles HR, Rood J, Barnett JB, Willett WC, Rimm EB, Bassett DR Jr. Physical Activity Assessment with the ActiGraph GT3X and Doubly Labeled Water. Med Sci Sports Exerc. 2017 Sep;49(9):1935-1944. doi: 10.1249/MSS.0000000000001299. PMID 28419028
- [Background] Bammann K, Thomson NK, Albrecht BM, Buchan DS, Easton C. Generation and validation of ActiGraph GT3X+ accelerometer cut-points for assessing physical activity intensity in older adults. The OUTDOOR ACTIVE validation study. PLoS One. 2021 Jun 3;16(6):e0252615. doi: 10.1371/journal.pone.0252615. eCollection 2021. PMID 34081715
- [Background] Aguilar-Farias N, Peeters GMEEG, Brychta RJ, Chen KY, Brown WJ. Comparing ActiGraph equations for estimating energy expenditure in older adults. J Sports Sci. 2019 Jan;37(2):188-195. doi: 10.1080/02640414.2018.1488437. Epub 2018 Jun 18. PMID 29912666
- [Derived] Zielinski OB, Hallager DW, Jensen KY, Carreon L, Andersen MO, Diederichsen LP, Bech RD. Multicentre investigation on the effect of decompressive surgery on Balance and physical ActiviTy Levels amongst patients with lumbar Spinal stenosis (B-ATLAS): protocol for a prospective cohort study. BMJ Open. 2024 Sep 23;14(9):e085667. doi: 10.1136/bmjopen-2024-085667. PMID 39313282